CLINICAL TRIAL: NCT02664090
Title: Hemodynamic Assessment With Trans-esophageal Doppler (TED) During Prone Ventilation in Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Hemodynamic Assessment With Trans-esophageal Doppler (TED) During Prone Ventilation in ARDS Patients
Status: Completed | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Mohan Gurjar, Associate Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2015-139-DM-88
Record Dates: First submitted 2016-01-15; First posted 2016-01-26 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: acute respiratory distress syndrome; prone ventilation; trans-esophageal doppler
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute respiratory distress syndrome (ARDS) commonly complicates acute illness in ICU. This syndrome is associated with high morbidity and mortality. In management of ARDS patients, lung protective ventilation and prone ventilation are key strategies which have shown survival benefits in recent years. Prone positioning has been reported to have hemodynamic disturbances like hypotension and arrhythmias. The literature till date is unclear with regards to acute hemodynamic changes which can happen during initiation of prone ventilation ,with a few studies suggesting decreasing cardiac output and a few increasing cardiac output. In recent years, trans-esophageal Doppler (TED) has become one of important hemodynamic assessment tool due to its minimal invasiveness, ease of use with its clinical utility established by various studies both in operation theatres and intensive care units. In current study, the investigators would like to evaluate acute hemodynamic effects of prone ventilation with TED in patients of acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
Introduction and rationale of the study:

Acute respiratory distress syndrome (ARDS) commonly complicates acute illness in intensive care units (ICU). This syndrome is associated with high morbidity and mortality. In management of ARDS patients, lung protective ventilation and prone ventilation are key strategies which have shown survival benefits in recent years and now becomes standard part of care in these patients. Prone positioning has been reported to have hemodynamic disturbances like hypotension and arrhythmias. Prone ventilation can have different cardiovascular effects with a few suggesting increased cardiac output and few decreased cardiac output with unclear literature till date with one recent study suggesting that patients who have preload reserve had increased cardiac output when compared to patients with no preload reserve.

In ICU, hemodynamic monitoring is being done as a part of standard care of management in critically ill patients. There are different modalities of continuous hemodynamic monitoring, which help in timely assessment and appropriate interventions to optimize cardiac output to maintain adequate organ perfusion in these critically ill patients. Cardiac output could be assessed by thermo-dilution technique with pulmonary artery catheter, pulse contour analysis of arterial waveform or echocardiography. In recent years, trans-esophageal Doppler (TED) has become one of the standard hemodynamic assessment tool in ICU due to its minimal invasiveness and easy to use. TED uses Doppler shift principle which is routinely used to measure cardiac output in both trans-thoracic and trans-oesophageal echocardiography. The clinical utility of TED, with the benefit of minimal invasiveness, in assessing hemodynamic perturbations in both operation theatre and ICU has been established by various studies. Doppler measured cardiac output showed high validity and clinical agreement with gold standard pulmonary artery thermo-dilution technique, which is more invasive. Hemodynamic assessment in prone position with TED has been studied intra-operatively with good correlation. In current study, the investigators will evaluate acute hemodynamic effects of prone ventilation with TED in patients of acute respiratory distress syndrome (ARDS).

Work plan methodology:

This will be a prospective, observational study, to be conducted in 12 bedded ICU of department of Critical Care Medicine, Sanjay Gandhi Institute of Postgraduate and Medical Sciences, Lucknow. Patients with ARDS whose hemodynamic monitoring is being done by TED, and planned for prone ventilation by treating physician's decision, will be screened for inclusion in this study.

After informed consent from patient's family member for inclusion in the study, demographic data including age, sex, weight, height and ideal body weight (IBW) will be noted. All study participants will have trans-thoracic echocardiography done before inclusion to exclude conditions that can interfere with oesophageal doppler readings like aortic coarctation, severe aortic stenosis, or severe aortic regurgitation. Hemodynamic monitoring with TED (Cardio Q) in these patients will be decided and initiated by treating clinician. As a part of standard treatment for ARDS, all patients will be receiving lung protective ventilation strategies as per ARDS net protocol with appropriate sedation, and also these patients will have relevant invasive and non-invasive vitals monitoring as per ICU protocol.

After decision for prone ventilation by treating clinician and obtaining consent for inclusion in this study, prior to any parameter measurement during study period, probe position of TED will be verified to ensure optimal acquisition of maximum velocity signal. Baseline hemodynamic and respiratory parameters (T1) will be noted in 45 degree head elevation position. Second set (T2) of hemodynamic parameters will be noted after passive leg raise test (PLR). Third set (T3) of hemodynamic parameters in supine position along with IAP measurement.

All ARDS patients will be proned as per ICU protocol, with protective measures for eyes, extended arms, and using appropriate thoraco-pelvic supports for unloading the abdomen and taking all other precautions required for prone positioning. After proning, transducers for invasive monitoring will be re-zeroed relative to atmospheric pressures.

Fourth set (T4) of parameters (hemodynamic) 5 minutes after prone ventilation will be noted. While, fifth set (T5) of parameters (hemodynamic, respiratory and IAP) will be noted 10 minutes after prone ventilation. Subsequently, hemodynamic parameters will be noted at 20 minutes (T6) and the last set (T7) of parameters (hemodynamic and respiratory) will be noted 30 minutes after initiation of prone ventilation.

Sample size calculation: Sample size was calculated by power analysis using PASS 2008 software, with difference in means of cardiac output of 0.6 litre/minute/meter2 between two paired groups and with 95% confidence interval (CI) and 80% power of the study, 22 patients will require. So, the investigators planned to include 25 patients for our study.

Data collection: Demographic and clinical characteristics (ventilatory and hemodynamics) of all included patients will be collected on structured proforma. ICU prognostication scores, i.e., Acute Physiologic and Chronic Health Evaluation (APACHE) II score and Sequential Organ Dysfunction Assessment (SOFA) will also be recorded. From baseline parameters noted before turning the patient prone and after PLR, hemodynamic, ventilatory parameters at sequential time intervals will be noted down until thirty minutes after initiation of prone ventilation.

Intervention: Nil. All patients will be managed as per the ICU treating team's decision

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years) with ARDS undergoing prone ventilation

Exclusion Criteria:

* Patients with age <18 years.
* Conditions which can interfere with interpretation of hemodynamic parameters through TED (aortic coarctation, severe aortic stenosis, severe aortic regurgitation, severe scoliosis)
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All critically ill adult patients with diagnosis of ARDS whose hemodynamic monitoring is being done by trans-esophageal doppler (TED), and planned for prone ventilation by treating physician's decision, will be screened for inclusion in this study.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
To measure pattern of changes in cardiac index (L/min/m2) from baseline (pre-prone position) to during prone position. | Baseline (pre-prone) and after initiation of prone-ventilation at 5, 10, 20 and 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Gurjar, MD, PDCC, Principal Investigator — Sanjay Gandhi Postgraduate Institute of Medical Sciences
Locations (1):
- Department of Critical Care Medicine, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Derived] Saran S, Gurjar M, Azim A, Mishra P, Ghosh PS, Baronia AK, Poddar B, Singh RK. Trans-Esophageal Doppler Assessment of Acute Hemodynamic Changes Due to Prone Positioning in Acute Respiratory Distress Syndrome Patients. Shock. 2019 Oct;52(4):e39-e44. doi: 10.1097/SHK.0000000000001290. PMID 30475331
- See also: Saran S, Gurjar M, Azim A, Mishra P, Ghosh PS, Baronia AK, et. al. Trans-Esophageal Doppler Assessment of Acute Hemodynamic Changes Due to Prone Positioning in Acute Respiratory Distress Syndrome Patients. Shock. 2019 Oct;52(4):e39-e44. PMID:30475331 — https://www.ncbi.nlm.nih.gov/pubmed/30475331